CLINICAL TRIAL: NCT03929822
Title: Contrast-Enhanced Spectral Mammography: Potential to Improve Diagnostic Accuracy
Brief Title: Can Contrast-Enhanced Spectral Mammography Improve the Accuracy of a Diagnosis
Status: Terminated | Type: Observational
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-116
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Breast Screening
Keywords: Mammography; Contrast-Enhanced Spectral Mammography; 19-116

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Contrast-Enhanced Spectral Mammography (CESM): Women called back from an abnormal screening mammogram/tomosynthesis exam will be offered CESM as part of their diagnostic work up. The radiologist will interpret the low energy images and record their findings.
  Interventions: Diagnostic Test: Contrast-Enhanced Spectral Mammography

INTERVENTIONS:
Diagnostic Test: Contrast-Enhanced Spectral Mammography — A standard dose of contrast material for other contrast mammography examinations and for body CT scanning, 1.5 ml/kg of Iohexol350 will be injected intravenously (IV) using a power injection (3-4 ml/s) with a maximum does of 150 ml. The IV injection is performed while the patient is in a sitting position. The mammogram will be performed in a standing position.

SUMMARY:
The purpose of this study is to test whether contrast-enhanced spectral mammography (CESM) may be able to reduce the number of unnecessary biopsies in women whose screening mammograms had abnormal findings.

ELIGIBILITY:
Inclusion Criteria:

* Women called back from a screening mammography by either FFDM or tomosynthesis with soft tissue abnormalities including masses, asymmetries, focal asymmetries or architectural distortion with or without calcifications. Patients will be questioned regarding the possibility of pregnancy and will need a negative pregnancy test prior the study intervention.

Exclusion Criteria:

* Age <30 years old
* Screening mammography with only calcifications abnormalities
* Male patients
* Pregnant or lactating patients
* Patients with any allergy to iodinated contrast
* Patients with eGFR < 45
* Patients that may be treated with radioactive iodine

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women called back from a screening mammography by either FFDM or tomosynthesis with soft tissue abnormalities including masses, asymmetries, focal asymmetries or architectural distortion with or without calcifications.
Study Population: Women called back from an abnormal screening mammogram/tomosynthesis exam will be offered CESM as part of their diagnostic work up.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of CESM compared to mammography | 2 years
  The radiologist will interpret the low energy images and record their findings.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Sung, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm